CLINICAL TRIAL: NCT06779578
Title: The Efficacy and Safety of Fluoroscopic-Guided Bipolar Versus Monopolar Pulsed Radiofrequency for Refractory Trigeminal Neuralgia: An Exploratory Study
Brief Title: Fluoroscopic-Guided Bipolar Versus Monopolar Pulsed Radiofrequency for Refractory Trigeminal Neuralgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Eman Hamdy, Lecturer in Neurology, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0307084
Record Dates: First submitted 2025-01-13; First posted 2025-01-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Trigeminal Neuralgia; Refractory Pain
Keywords: trigeminal neuralgia; Radiofrequency ablation; Pulsed radiofrequency; Monopolar pulsed radiofrequency; Bipolar pulsed radiofrequnency
MeSH Terms: conditions — Trigeminal Neuralgia; Pain, Intractable

STUDY DESIGN:
Intervention Model Description: Explaratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Monopolar pulsed radiofrequncy (Placebo Comparator): Patients with refractory TN undergoing monopolar pulsed radiofrequency
  Interventions: Procedure: Mopolar pulsed radiofrequency
- Bipolar pulsed radiofrequency (Active Comparator): Patients with refractory TN undergoing bipolar pulsed radiofrequency
  Interventions: Procedure: Bipolar pulsed radiofrequency

INTERVENTIONS:
Procedure: Bipolar pulsed radiofrequency — Bipolar pulsed radiofrequency ablation: the active comparator
  Arms: Bipolar pulsed radiofrequency
Procedure: Mopolar pulsed radiofrequency — Monopolar pulsed radiofrequency ablation: the placebo
  Arms: Monopolar pulsed radiofrequncy

SUMMARY:
A prospective exploratory study aiming at comparing pulsed bipolar versus pulsed unipolar radiofrequency ablation in patients with medically refractory trigeminal neuralgia.

DETAILED DESCRIPTION:
This will be a prospective exploratory that will be conducted on patients with the inclusion and exclusion criteria detailed.

At the baseline visit, the sociodemographic data (age, sex, smoking status) and clinical data (TN etiology (idiopathic or symptomatic), TN phenotype (purely paroxysmal or with concomitant continuous pain), clinical symptoms topography (V2, V3), brain MRI findings, previous medications and interventions, and comorbidities) will be collected. The patients will be randomly assigned to undergo bipolar PRF or monopolar PRF using a simple randomization technique.

Pain scores will be assessed using the nominal rating scale (NRS) at baseline, within two weeks postoperatively, and at 1-month, 3-month, and 6-month intervals. Patient satisfaction will be assessed within two weeks following the intervention on a five-point Likert scale (5 represents very good and 1 means very bad). Treatment success will be defined as at least a 50% reduction in pain scores. The duration to pain control and the duration to pain recurrence/rebound will be assessed at follow-up visits. The patient's postoperative need for medications or further pain interventions will be detailed. Intraoperative and postinterventional complications will be monitored and documented.

Study interventions For the PRF procedure, all patients will be prepared in the operating room and will undergo standard operative monitoring (i.e., blood pressure, electrocardiography, and pulse oximetry). They will be positioned in a supine position with slight neck extension. Sedation will be provided (100 Ig fentanyl and 2 mg midazolam intravenously). Skin preparation will be performed using chlorhexidine.

I- Monopolar PRF In the monopolar PRF, an RF cannula (22-gauge, 100 mm, with a 10 mm active tip (SMK)) will be percutaneously advanced at the posterior border of the foramen ovale under fluoroscopic guidance. For confirming the detection of the mandibular nerve, sensory stimulation will be performed via the radiofrequency generator at a current of 0.5 to 1 V at a frequency of 50 Hz to elicit paresthesia response in the mandibular region. Motor stimulation will be performed via the generator at a current of 1 - 2 V applied at a frequency of 2 Hz to obtain a contraction response at the masseter muscle. After obtaining the appropriate responses, PRF will be applied at a fixed heat energy of 42 °C for a period of 240 seconds10.

II- Bipolar PRF For bipolar PRF, two RF cannulas will be advanced in the foramen ovale under fluoroscopic guidance. The first (22-gauge, 100 mm, and 10-mm active tip (SMK)) will be placed at the anterior border of the foramen ovale, and then the second (same parameters) will be advanced at the posterior border. The correct position will be confirmed on the lateral position until the correct placement at V2. Sensory and motor testing will be performed as aforementioned in the monopolar PRF to confirm the appropriate capture of the trigeminal nerve. Following obtaining the appropriate responses, PRF will be performed in two cycles, three minutes each, at a temperature of 42ºC and a current of 85 V and a 20-millisecond pulse width13.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a definitive diagnosis of classical TN based on the third version of the International Classification of Headache Disorders (ICHD-3).
2. Either purely paroxysmal classical TN or classical TN with concomitant chronic pain.
3. Patients with idiopathic TN, with symptomatic clinical topography of V2 and/or V3.
4. Patients with brain magnetic resonance imaging (MRI) unremarkable for structural etiology for the trigeminal pain.
5. Patients with medically refractory TN defined as pain persisting beyond three months at a level of ≥5/10 after monotherapy or polytherapy in appropriate medical doses.

Exclusion Criteria:

1. Painful trigeminal neuropathy based on the third version of the International Classification of Headache Disorders (ICHD-3).
2. Trigeminal neuralgia with V1 symptomatic clinical topography.
3. Trigeminal neuralgia comorbid with other atypical facial pain disorders.
4. Structural TN e.g., due to vascular compression, posterior fossa tumors, central demyelination, …etc.
5. Patients exposed to previous radiofrequency procedures, as this may impair the nerve response to current PRF.
6. Patients who refused to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Numerical pain scale (NRS) | Two weeks, 1 month, 3 months, and 6 months
  50% Pain reduction in the numerical rating scale (NRS)

SECONDARY OUTCOMES:
Adverse events monitoring (Frequency, severity, seriousness, and causality) | 6 months
  Frequency, type, and severity of adverse events. Classification of AEs as mild, moderate, or severe. Assessment of causality between the treatment and the AE

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Alexandria University Faculty of Medicine, Alexandria
  - Cairo University Kasr Alainy Faculty of Medicine, Cairo

IPD SHARING:
Plan to Share IPD: Undecided